CLINICAL TRIAL: NCT06619132
Title: Training Load Adapted to Muscle Properties to Reduce Injury Occurrence in Sprint
Acronym: FULGUR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French National Insitute of Sport (Unknown); FULGUR consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-A02523-38; ANR-19-STHP-0003 (Other: ANR)
Record Dates: First submitted 2024-08-23; First posted 2024-10-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: NON APPLICABLE
Keywords: Sprint; Performance; High elite athletes; injury; hamstring
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
During the Olympics, running fast is the most prevalent motor task, 100-m dash being the one of the most-expected event. Yet, the achievement of such running sprints requires both extreme athletic capabilities together with robust musculoskeletal system in order to limit the risk of injury. Lower limb muscle injury is indeed the main cause of training or competition interruption on the international stage. In this context, France presents the unique feature of being historically strong in velocity-oriented sports and recognized for the quality of research work done for the understanding of sprint running performance. This research program will be conducted in strong collaboration with French Federations of Athletics, Rugby and Ice Sports (bobsleigh). FULGUR gathers world's leading experts in muscle biomechanics, strength and conditioning research, clinical imaging, health behaviors, and machine learning applied to very high sport performance in order to pursue a threefold objective:

* To appraise sprint mechanics at center of mass and joint segments level in a view to quantify specific-structure workload at these scales in ecological conditions (Workpackage 1);
* To determine individual musculoskeletal profile of elite athlete to propose tailored strengthening programs in order to optimize running propulsion efficiency (Workpackage 2);
* To estimate the level of injury risk and suggest individualized prevention contents based on a multi-factorial approach (Workpackage 3).

These goals will be supported by transverse tasks aiming at refining muscle mechanics and motion capture analysis based on ultrasound imaging and machine learning. These tasks will aim to advance the analysis of skeletal muscle dynamics 2D ultrasound analyses and to implement markerless motion capture methods in the field. Led by the flagship French laboratory focused on very high sport performance, these work originate from long-term collaborations between high-end athletic and multi-disciplinary scientific staffs. Thanks to a strong evidence-based methodological approach and minimal time-cost for top-level athletes, all the efforts put in FULGUR will convert to the ultimate goal of fast-track knowledge and tech transfer towards sport performance stakeholders. Tailored-made sprint, strength and prevention training will be co-built with coaches and staffs during panel meetings in a view to optimize sprint performance and reduce the exposure of top-level French sprinters, rugby 7 players and bobbers to muscle injury. The knowledge inferred from this project will have direct implications in every discipline that elicits all-out sprints and accelerations (e.g. team sports, racket sports). Regular meetings with coaches and heads of federal R&D departments will result in a strongly anticipated strategy to enhance the potential of knowledge transfer and performance optimization (annual expertise meetings, innovative videos including dynamic infographics, short technical sheets, expert education programs for coaches). This approach is expected to strongly contribute to upgrade scientific skills of French performance stakeholders from Tokyo 2020 to Paris 2024 and beyond.

DETAILED DESCRIPTION:
During the Olympics, running fast is the most prevalent motor task, 100-m dash being the one of the most-expected event. Yet, the achievement of such running sprints requires both extreme athletic capabilities together with robust musculoskeletal system in order to limit the risk of injury. Lower limb muscle injury is indeed the main cause of training or competition interruption on the international stage. In this context, France presents the unique feature of being historically strong in velocity-oriented sports and recognized for the quality of research work done for the understanding of sprint running performance. This research program will be conducted in strong collaboration with French Federations of Athletics, Rugby and Ice Sports (bobsleigh). FULGUR gathers world's leading experts in muscle biomechanics, strength and conditioning research, clinical imaging, health behaviors, and machine learning applied to very high sport performance in order to pursue a threefold objective:

* To appraise sprint mechanics at center of mass and joint segments level in a view to quantify specific-structure workload at these scales in ecological conditions (Workpackage 1);
* To determine individual musculoskeletal profile of elite athlete to propose tailored strengthening programs in order to optimize running propulsion efficiency (Workpackage 2);
* To estimate the level of injury risk and suggest individualized prevention contents based on a multi-factorial approach (Workpackage 3).

These goals will be supported by transverse tasks aiming at refining muscle mechanics and motion capture analysis based on ultrasound imaging and machine learning. These tasks will aim to advance the analysis of skeletal muscle dynamics 2D ultrasound analyses and to implement markerless motion capture methods in the field. Led by the flagship French laboratory focused on very high sport performance, these work originate from long-term collaborations between high-end athletic and multi-disciplinary scientific staffs. Thanks to a strong evidence-based methodological approach and minimal time-cost for top-level athletes, all the efforts put in FULGUR will convert to the ultimate goal of fast-track knowledge and tech transfer towards sport performance stakeholders. Tailored-made sprint, strength and prevention training will be co-built with coaches and staffs during panel meetings in a view to optimize sprint performance and reduce the exposure of top-level French sprinters, rugby 7 players and bobbers to muscle injury. The knowledge inferred from this project will have direct implications in every discipline that elicits all-out sprints and accelerations (e.g. team sports, racket sports). Regular meetings with coaches and heads of federal R&D departments will result in a strongly anticipated strategy to enhance the potential of knowledge transfer and performance optimization (annual expertise meetings, innovative videos including dynamic infographics, short technical sheets, expert education programs for coaches). This approach is expected to strongly contribute to upgrade scientific skills of French performance stakeholders from Tokyo 2020 to Paris 2024 and beyond.

ELIGIBILITY:
Inclusion Criteria:

* French high elite athlete form athletics, rugby 7 and bobsleigh

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: French high elite athlete form athletics, rugby 7 and bobsleigh
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Sprint power and performance | through study completion, an average of 4 years
  Force-power-velocity profile during a maximal free sprint

SECONDARY OUTCOMES:
Musculo-skeletal characteristics, training load, psychological characteristics | through study completion, an average of 4 years
  Musculo-skeletal characteristics : joint force, power, velocity at the hip, knee and ankle level (isokinetic testing), muscle elasticity (ultra sound elastography), muscle architecture and geometry (ultrasound, MRI), muscle coordination (EMG) Training load (RPE, GPS quatification)
Psychological characteristics evaluation | through study completion, an average of 4 years
  A measurement tool established by our study team will be used to assess the measure, named: For anxiety, motivation, optimism, impulsivity, emotion self regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Gaël GUILHEM, PhD, Principal Investigator — Laboratory of sport, expertise and performance - National Institut of Sport of Expertise and Performance
Locations (1):
- French National Insitute of Sport, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edouard P, Caumeil B, Verhagen E, Guilhem G, Ruffault A. Maximising individualisation of sports injury risk reduction approach to reach success. Braz J Phys Ther. 2022 May-Jun;26(3):100394. doi: 10.1016/j.bjpt.2022.100394. Epub 2022 Feb 12. PMID 35526371
- [Background] Fornasier-Santos C, Arnould A, Jusseaume J, Millot B, Guilhem G, Couturier A, Samozino P, Slawinski J, Morin JB. Sprint Acceleration Mechanical Outputs Derived from Position- or Velocity-Time Data: A Multi-System Comparison Study. Sensors (Basel). 2022 Nov 8;22(22):8610. doi: 10.3390/s22228610. PMID 36433206
- See also: https://www.enseignementsup-recherche.gouv.fr/fr/le-sprint-vaste-programme-de-recherche-avec-fulgur-96045 — https://labos-recherche.insep.fr/fr/laboratoire-sep/fulgur